CLINICAL TRIAL: NCT01537952
Title: Microbiologic Findings of Acute Facial Palsy in Children
Status: Completed | Type: Observational
Sponsor: University of Helsinki (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Mervi Kanerva, MD, PhD, University of Helsinki
Other Study IDs: 230419
Record Dates: First submitted 2012-02-18; First posted 2012-02-23 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Facial Paralysis
Keywords: facial paralysis, facial nerve, borreliosis, Bell's palsy
MeSH Terms: conditions — Facial Paralysis; Borrelia Infections; Bell Palsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective: Microbiologic etiologies of facial palsy in children were investigated.

Study design: Prospective clinical study. Methods: Forty-six children aged 0-16 years with facial palsy comprised the study group. Paired serum samples and cerebrospinal fluid were tested to find indications (antibodies, growth of the microbe, or nucleic acids) of microbes putatively associated with facial palsy. The microbes tested were herpes simplex virus-1 and -2, varicella-zoster virus, human herpesvirus-6, Mycoplasma pneumoniae, Borrelia burgdorferi, influenza A and B-, picorna-, cytomegalo-, parainfluenza-, respiratory syncytial-, coxsackie B5-, adeno-, and enteroviruses, Chlamydia psittaci, and Toxoplasma gondii. Besides the routine tests in clinical practice, serum and cerebrospinal fluid samples were tested with a highly sensitive microarray assay for DNA of herpes simplex virus-1 and -2, human herpesvirus-6A , -6B, -7, Epstein-Barr-, cytomegalo-, and varicella-zoster viruses.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-16
* Facial palsy

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Tertiary university Hospital, children 0-16 years old
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2007-05; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

REFERENCES:
- [Derived] Kanerva M, Nissinen J, Moilanen K, Maki M, Lahdenne P, Pitkaranta A. Microbiologic findings in acute facial palsy in children. Otol Neurotol. 2013 Sep;34(7):e82-7. doi: 10.1097/MAO.0b013e318289844c. PMID 23657208